CLINICAL TRIAL: NCT03211871
Title: Dexmedetomidine Infusion as an Analgesic Adjuvant During Laparoscopic Cholecystectomy: Randomized Controlled Study
Brief Title: Dexmedetomidine Infusion as an Analgesic Adjuvant During Laparoscopic Cholecystectomy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bogomolets National Medical University (Other)
Responsible Party: Principal Investigator, Kateryna Bielka, assistant professor at Anesthesiology and intensive care Department, Bogomolets National Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 87678
Record Dates: First submitted 2017-07-04; First posted 2017-07-07 (Actual); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Pain, Postoperative
Keywords: pain management, dexmedetomidine
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: After the primary patient assessment, eligible participants were assigned in a 1:1 ratio to either the intervention (Group D) or control (Group C) groups using random assignment in blocks of four.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group D (Active Comparator): Group D received dexmedetomidine infusion 0,5 mcg/kg/h from induction in anesthesia to extubation
  Interventions: Drug: Dexmedetomidine
- Croup C (Placebo Comparator): group C (control) received normal saline infusion
  Interventions: Drug: Normal Saline Flush, 0.9% Injectable Solution_#1

INTERVENTIONS:
Drug: Dexmedetomidine — Intraoperative intravenous dexmedetomidine infusion 0,5 mcg/kg/h
  Arms: Group D
Drug: Normal Saline Flush, 0.9% Injectable Solution_#1 — Intraoperative intravenous normal saline infusion
  Arms: Croup C

SUMMARY:
The aim of this study was to evaluate efficacy and safety of dexmedetomidine infusion during laparoscopic cholecystectomy. The randomized, single-center, controlled study was carried out from May 2016 to June 2017 at department of surgery, anesthesiology and intensive care, Postgraduate Institute of Bogomolets National Medical University.

DETAILED DESCRIPTION:
Dexmedetomidine provide sedative, sympatholytic and analgesic effect, so it could be used as an adjuvant to improve analgesia, hemodynamic response to intubation and pneumoperitoneum, decrease the number of opioid-associated adverse effects.

The aim of this study was to evaluate efficacy and safety of dexmedetomidine infusion during laparoscopic cholecystectomy.

The randomized, single-center, controlled study was carried out from May 2016 to June 2017 at department of surgery, anesthesiology and intensive care, Postgraduate Institute of Bogomolets National Medical University. Study design was approved by Ethical Committee at Bogomolets National Medical University (approval code 56).

60 patients elected for LCE were included in the study. The inclusion criteria were: age between 18 and 79 years, either sex, American Society of Anesthesiology (ASA) physical status I to II. The exclusion criteria were age outside the specified range, pregnancy or lactation, severe systemic disease (ASA III physical status), patients on b-blockers or calcium channel blockers.

After the primary patient assessment, eligible participants were assigned in a 1:1 ratio to either the intervention (Group D) or control (Group C) groups using random assignment in blocks of four. The randomization sequence was generated using a computer algorithm [19]. Randomization and data analysis were conducted by an independent blinded member of the research team.

Group D received dexmedetomidine infusion 0,5 mcg/kg/h from induction in anesthesia to extubation, group C (control) received normal saline infusion. To prepare the infusion, dexmedetomidine 2ml containing 100mcg of the drug was diluted up to 50 ml with normal saline resulting in final concentration of 4mcg/kg. Dexmedetomidine or normal saline infusion was given through infusion pump.

After taking the patient to the operation room, vital signs monitor Philips and Bispectral Index (BIS) monitoring were attached (pulse, heart rate, electrocardiography (ECG), arterial pressure (AP), oxygen saturation). Peripheral intravenous cannula was inserted for intravenous fluids and infusion pump (separate line). Patients did not receive premedication. Before induction they receive dexketoprofen 50mg IV and omeprazole 40mg.

Pre-oxygenation was performed for 2 min, induction in anesthesia - with propofol 2mg/kg IV and succinyl choline 1,5mg/kg IV. After intubation anesthesia was maintained with sevoflurane and atracurium bromide. The patients were ventilated with circle system with goal CO2 35-45 mm Hg. BIS-monitor target was between 40 and 60. Anesthetics and drug infusion were stopped with the end of surgery.

The primary efficacy outcomes were number of patients with severe pain, time to first rescue analgesia and postoperative morphine consumption. Severe pain was estimated as VAS≥7 during 30% or more time in first 48 hours after surgery. Time to first rescue analgesia was estimated as time from end of anesthesia to the time postoperatively when patient ask for analgesia or have VAS≥4. Injection morphine hydrochlorides 10mg subcutaneously was used as a rescue analgesic. NSAIDs (dexketoprofen 150mg per day) were prescribed routinely.

Secondary efficacy outcomes included:

* Time from end of surgery to extubation
* Lengths of postanesthesia unit/general ward stay
* Incidence of chronic postoperative pain During first 48 hours after surgery patients in both groups were evaluated by the nursing stuff using the Richmond agitation sedation scale (RASS) for sedation, visual analogue scale (VAS) for pain assessment (every 2 hours or prior to rescue analgesia).

Safety was assessed by monitoring vital signs and recording adverse events. During anesthesia all patients receive continuous ECG, BIS, pulse oximetry, capnography monitoring. AP was measured every 3-5min. Arterial blood gases were checked by doctor prescription. An adverse event was recorded if systolic blood pressure was <90 or >160 mmHg or if heart rate was <50 or >110 beats/min; desaturation was estimated as peripheral oxygen saturation (or SaO2) <90%. Interventions for bradycardia, tachycardia, hypertension and hypotension comprised titration or interruption of study agent, or additional drug therapy.

Statistical analysis was performed using R software. Categorical data are presented as proportions and continuous data as medians with 25-75% interquartile ranges (IQRs). Chi-square testing demonstrated that all of the study variables were discrete. To assess significance levels, a two-tailed Mann-Whitney U-test and Fisher's exact test were used. A p-value of <0.05 was considered significant.

ELIGIBILITY:
Inclusion Criteria:

* patients elected for laparoscopic cholecystectomy
* age between 18 and 79 years
* either sex
* ASA physical status I to II

Exclusion Criteria:

* age outside the specified range
* pregnancy or lactation
* severe systemic disease (ASA III physical status or more)
* patients on b-blockers or calcium channel blockers

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-05-01 (Actual); Primary Completion 2017-08-01 (Estimated); Study Completion 2017-10-01 (Estimated)

PRIMARY OUTCOMES:
number of patients with severe pain | 48 hours after surgery
  number of patients with severe pain estimated as VAS≥7 during 30% or more time in first 48 hours after surgery
Time to first rescue analgesia | 24 hours after surgery
  time from end of anesthesia to the time postoperatively when patient ask for analgesia or have VAS≥4
morphine consumption | 48 hours
  total morphine consumption after surgery in mg

SECONDARY OUTCOMES:
Time of extubation | 24 hours after surgery
  Time from end of surgery to extubation
Incidence of chronic postoperative pain | 6 month after surgery
  number of patients with chronic postoperative pain

CONTACTS AND LOCATIONS:
Locations (1):
- Kyiv Clinical City Hospital #1, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: Undecided
IPD will not be available

REFERENCES:
- [Derived] Bielka K, Kuchyn I, Babych V, Martycshenko K, Inozemtsev O. Dexmedetomidine infusion as an analgesic adjuvant during laparoscopic small es, Cyrillicholecystectomy: a randomized controlled study. BMC Anesthesiol. 2018 Apr 20;18(1):44. doi: 10.1186/s12871-018-0508-6. PMID 29678158